CLINICAL TRIAL: NCT00339469
Title: The Effects of a High Legume Low Glycemic Index Diet on Insulin Resistance and Inflammation in Patients at High Risk for Colorectal Adenoma Recurrence
Brief Title: Effect of High-Legume Diet on Colorectal Cancer Risk
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 999905215; 05-C-N215; NCT00557063 (obsolete NCT alias)
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2018-02-13

CONDITIONS: Inflammation; Prevention and Control; Colonic Neoplasms; Diet; Insulin
Keywords: Prevention; Colorectal Neoplasms; Insulin Resistance; Inflammation Obesity; Adenoma
MeSH Terms: conditions — Inflammation; Colonic Neoplasms; Insulin Resistance; Colorectal Neoplasms; Adenoma

ARMS (1):
- 2 (Other): Controlled feeding study.
  Interventions: Dietary Supplement: LIFE

INTERVENTIONS:
Dietary Supplement: LIFE — We are evaluating the effects of a legume enriched, low glycemic index, high fermentable fiber diet, on CRP, and C-peptide participants with four possible combinations of the risk factors insulin resistance and history of adenomatous polyps. In a randomized crossover design controlled feeding study each participant consumed the above experimental diet and a control diet for four weeks with a two week washout period between diets. 65 male participants were recruited and randomized into four groups. A secondary objective is to assess whether these endpoints change by IR status or a history of adenomas. In addition, potential fecal markers of CRC risk are being measured to assess changes in gastrointestinal inflammation, including mRNA from exfoliated fecal colonocytes. To our knowledge this is the first controlled feeding study: 1. to examine the effects of legumes or a low GI diet on markers of inflammation

SUMMARY:
This study, sponsored by the National Cancer Institute and Penn State University, will examine how a diet high in legumes (dried beans) influences risk factors for colon cancer and polyps. Many scientists believe that colon and rectal cancers develop from polyps (tumors of the lining of the large bowel). This study will test whether a high-legume diet can reduce levels of certain factors (blood insulin, blood glucose, and markers of inflammation such as C-reactive protein) that at elevated levels are known to increase the risk of colorectal polyps and colon cancer.

Healthy men between 35 and 75 years of age may be eligible for this study, conducted at Penn State University in University Park, Pennsylvania. Candidates are screened with blood tests and measurements of height, weight, and blood pressure. All candidates must have had a colonoscopy within 2 years of entering the study. They may or may not have had adenomas and may or may not be insulin-resistant. Candidates must not have cancer, heart disease, kidney disease, diabetes, or other serious medical condition, and they must have no history of colorectal cancer, polyp removal, bowel surgery, polyposis syndrome, or inflammatory bowel disease. Participants undergo the following tests and procedures:

* Caloric requirement testing: The subject's resting metabolic rate is measured while fasting and in the early morning at rest to determine daily calorie requirement before beginning the study diet. A special clear plastic hood is placed over the subject's head while his breathing is measured. He can communicate with the technician at all times during the 30-minute test.
* Study diet: Subjects follow two required 4-week diets with a 3-week break in between, followed by an optional third 4-week diet. Subjects eat a healthy American diet for both of the required 4-week diet periods; about 1-1/2 cups of cooked legumes, such as pinto, baked, and navy beans are added to one of the two required diets. For the third (optional) diet period, subjects are given the same 1-1/2 cups of legumes, but are allowed to lose weight. Participants are given packages with all of the food they are to consume during the three diet periods. They may add up to five caffeine-containing beverages per day and up to two alcoholic drinks per week. They must eat all of the food they are given and only the food they are given. Subjects are expected to maintain a constant body weight during the two 4-week required diets, and their caloric intake may be increased or decreased as needed to maintain their screening weight.
* Weight measurements: Subjects are weighed regularly at the clinic.
* Blood samples: Subjects have blood samples drawn at the mid-point of each of the two required 4-week diets and at the beginning and end of each of the three 4-week diets.
* Urine and stool samples: Urine and stool samples are collected at the beginning and end of the two required 4-week diets.

DETAILED DESCRIPTION:
Clinical, epidemiological, and molecular studies provide compelling evidence that most colorectal cancers arise from adenomas. The epidemiology of adenomas closely resembles that of colorectal cancer itself, and prevention of adenomas will most likely prevent colorectal cancer. Insulin resistance and type 2 diabetes are emerging as significant risk factors for colorectal (CRC) cancer and adenomas. Insulin resistance is defined as impaired biological response to the action of insulin. It is characterized by compensatory hyperinsulinemia and is associated with increased risk for Type 2 diabetes. C-peptide, a marker of insulin production, is elevated in IR and is also a risk factor for CRC. Both insulin resistance and colorectal cancer are increasingly recognized as chronic, low-level, inflammatory states. C-reactive protein (CRP), an acute phase protein and a sensitive marker of sub-clinical inflammation, is a risk factor for both IR and CRC.

Analysis from the Polyp Prevention Trial (PPT), a multi-center, randomized trial of 1905 participants who had a colorectal adenoma, showed that legume consumption was significantly associated with reduction of both adenoma recurrence and advanced adenoma recurrence. Legumes are a rich source of dietary fibers and anti-inflammatory, anti-cancer phytochemicals.

We are evaluating the effects of a legume enriched, low glycemic index, high fermentable fiber diet, on CRP, (a measure of inflammation) and C-peptide (a measure of insulin resistance) in participants with four possible combinations of the risk factors insulin resistance and history of adenomatous polyps. In a randomized crossover design controlled feeding study each participant consumed the above experimental diet and a control diet for four weeks with a two week washout period between diets. 65 male participants were recruited and randomized into four groups. A secondary objective is to assess whether these endpoints change by IR status or a history of adenomas. In addition, potential fecal markers of CRC risk are being measured to assess changes in gastrointestinal inflammation, including mRNA from exfoliated fecal colonocytes. To our knowledge this is the first controlled feeding study: 1. to examine the effects of legumes or a low GI diet on markers of inflammation; 2. to compare the effects of a dietary intervention on patients with a history of colon adenomas with or without IR; and 3. to measure the effects of dietary changes in human intestinal gene expression profiles using exfoliated colonocytes.

ELIGIBILITY:
* INCLUSION CRITERIA

  1. Subjects are between 35-75 years old.
  2. Subjects are male.
  3. Subjects have a BMI 25.0-34.9 kg/m(2)

     Group 1 (adenoma, IR)
  4. Subjects had a colonoscopy within the last two years
  5. Subjects who had had one or more histologically confirmed adenomas removed from the colon during a colonoscopy in the last two years, in which the cecum was visualized, all polyps were removed, and the bowel was adequately prepared.
  6. Subjects have had either an adenoma previous to the above colonoscopy or multiple adenomas during the above colonoscopy.
  7. Subjects should have more than one previous adenoma in the colon. Rectal adenomas will be excluded. (If a person has only rectal adenomas or 1 colon and numerous rectal adenomas they will be excluded from the study, since the epidemiology for rectal and colon adenomas differ)
  8. Subjects are insulin resistance as determined by the Homeostasis Assessment Model (HOMA-IR), a mathematical model which allows values for insulin sensitivity and beta-cell function (expressed as percent of normal) to be obtained from simultaneous fasting plasma glucose and fasting insulin. HOMA-IRA is calculated by fasting serum insulin (FI in uU/mL); fasting glucose (FG in mmol/L) / 22.5 or HOMA-IR = FIxFG/22.5 (188). Values greater than or equal to 2.61 are considered insulin resistant

     Group 2 (adenomas, non IR)
  9. Subjects had a colonoscopy within the last two years.
  10. Subjects had one or more histologically confirmed colorectal adenomas removed during a colonoscopy in the last two years in which the cecum was visualized, all polyps were removed, and the bowel was adequately prepared.
  11. Subjects have had either an adenoma previous to the above colonoscopy or multiple adenomas during the above colonoscopy.
  12. Subjects should have more than 1 adenoma in the colon (vs rectum).
  13. Subjects are not insulin resistance as determined by HOMA-IR.

      Group 3 (no adenoma, IR)
  14. Subjects (controls) had a colonoscopy within the last two years and who had no histologically confirmed colorectal adenomas during the colonoscopy, in which the cecum was visualized and the bowel was adequately prepared.
  15. Subjects have had no previous adenoma.
  16. Subjects are insulin resistant as determine by HOMA-IR.

      Group 4 (no adenoma, non IR)
  17. Subjects (controls) had a colonoscopy within the last two years and had no histologically confirmed colorectal adenomas during the colonoscopy, in which the cecum was visualized and the bowel was adequately prepared.
  18. Subjects have had no previous adenomas.
  19. Subjects are not insulin resistance as determined by HOMA-IR.

EXCLUSION CRITERIA

All Subjects

1. A serious medical condition such as cancer, heart disease, kidney disease, diabetes or other serious medical condition.
2. A history of colorectal cancer, surgical resection of adenomas, bowel resection, the polyposis syndrome, or inflammatory bowel disease.
3. Smoked regularly in the past year.
4. Have a medical condition or dietary restrictions or practices that would substantially limit compliance with the dietary protocol.
5. Planning on changing diet, exercise or other health behavior in the next 6 months.
6. Taking any medication that may alter inflammation markers, insulin, glucose, and lipids.

Potential participants should not be regularly using the following preparations:

* Antibiotics
* Non-steroidal anti-inflammatory drugs (aspirin and other non-aspirin NSAIDS like inbuprofen, naproxen, indomethacin, piroxicam, COX-2-specific inhibitor drugs such as celecoxib, etodolac, and meloxicam)
* Glucocorticoids and other steroids
* Oral glucose preparations (e.g. Actos, Amaryl, Avandia, DiaBeta, Diabinese, Dymelor, Glucophage(XR), Glucotrol(XL), Glucovance, Glynase Pres Tab, Glyset, Micronase, Orinase, Prandin, Precose, Starlix, Tolinase)
* Insulin injections
* Statins (e.g. atorvastatin, fluvastatin, lovastatin, pravastatin, rosuvastatin, simvastatin)
* Bile Acid Resins (e.g. cholestyramine, colestipol, colesevelam)
* Nicotinic Acid (Niacin)
* Fibrates (e.g. clofibrate, fenofibrate, gemfibrozil)
* Combination Lipid Lowering Drugs (e.g. Crestor)

Participants will be asked not to use any supplements (including herbal and alternative therapies) other than a regular multi-vitamin/mineral while participating in the study. While we ask subjects to stop use of OTC medications during the study, we recognize that there may be occasional use of OTC analgesics during the course of the study. At least under some circumstances we will permit the use of OTC analgesics, which is otherwise listed as an exclusion criteria. At their scheduled blood draws, we will ask subjects to report any use of OTC medications during the past week. Participants will also be asked to limit their use of alcohol during the study to less than or equal to 2 drinks/week.

Ages: 35 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2005-08-03; Primary Completion 2008-05-19 (Actual); Study Completion 2018-02-13 (Actual)

PRIMARY OUTCOMES:
Biomarkers of insulin resistance and inflammation | At 6 weeks (end of study period)

SECONDARY OUTCOMES:
Weight loss | At 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Young, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Pennsylvania State University, University Park, Pennsylvania, United States

REFERENCES:
- [Background] Zhao C, Ivanov I, Dougherty ER, Hartman TJ, Lanza E, Bobe G, Colburn NH, Lupton JR, Davidson LA, Chapkin RS. Noninvasive detection of candidate molecular biomarkers in subjects with a history of insulin resistance and colorectal adenomas. Cancer Prev Res (Phila). 2009 Jun;2(6):590-7. doi: 10.1158/1940-6207.CAPR-08-0233. Epub 2009 May 26. PMID 19470793
- [Background] Hartman TJ, Albert PS, Zhang Z, Bagshaw D, Kris-Etherton PM, Ulbrecht J, Miller CK, Bobe G, Colburn NH, Lanza E. Consumption of a legume-enriched, low-glycemic index diet is associated with biomarkers of insulin resistance and inflammation among men at risk for colorectal cancer. J Nutr. 2010 Jan;140(1):60-7. doi: 10.3945/jn.109.114249. Epub 2009 Nov 4. PMID 19889807
- [Background] Zhang Z, Lanza E, Kris-Etherton PM, Colburn NH, Bagshaw D, Rovine MJ, Ulbrecht JS, Bobe G, Chapkin RS, Hartman TJ. A high legume low glycemic index diet improves serum lipid profiles in men. Lipids. 2010 Sep;45(9):765-75. doi: 10.1007/s11745-010-3463-7. Epub 2010 Aug 24. PMID 20734238